CLINICAL TRIAL: NCT07333053
Title: FOLFOX-Based Transarterial Infusion Chemotherapy for Unresectable Colorectal Cancer: An Open-Label, Multicenter, Randomized, Controlled, Phase Ⅱ Trial
Brief Title: Clinical Efficacy of Transarterial Infusion Chemotherapy for Unresectable Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quanda Liu (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other); The Rocket Force Characteristic Medical Center (Unknown); Second Affiliated Hospital of Nanchang University (Other); The Affiliated Hospital of Hebei University (Unknown); The First Hospital of Qinhuangdao (Other Government); The Central Hospital of Handan City (Unknown); The First People's Hospital of Jiujiang City (Unknown); Changzhi Medical College (Other); Zibo Boshan District Traditional Chinese Medicine Hospital (Unknown); Linshu County People's Hospital (Unknown); Hebei Yixian Hospital (Unknown); Baoding Mancheng District People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Quanda Liu, Chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-268-KY
Record Dates: First submitted 2025-12-18; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Unresectable Colorectal Cancer
Keywords: Transarterial Infusion Chemotherapy; Bevacizumab; Cetuximab; Colorectal Cancer; FOLFOX Protocol; Unresectable; Clinical Trial
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAIC Group (Experimental): Patients in the TAIC group will undergo FOLFOX-based TAIC combined with either cetuximab or bevacizumab on weeks 0 and 4, and will receive FOLFOX-based IVC combined with either cetuximab or bevacizumab on weeks 2 and 6. During each TAIC, based on the tumor's vaIVCular supply, the Seldinger technique is used to puncture the right femoral artery, and a microcatheter is inserted into the arterial branch of the superior mesenteric artery, inferior mesenteric artery, or common iliac artery, which is predominantly feeding the tumor. Chemotherapy drugs will be administered via the microcatheter. The FOLFOX-based TAIC consists of oxaliplatin (85 mg/m²) administered as a 2 hours transarterial infusion, leucovorin (400 mg/m²) administered as a 2 hours transarterial infusion, and fluorouracil (2400 mg/m²) administered as a 44 hours transarterial infusion, followed by intravenous administration of bevacizumab (5 mg/kg) or cetuximab (500 mg/m²). The IVC regimen is the same as that in the IVC group
  Interventions: Procedure: Transarterial infusion chemotherapy (TAIC)
- IVC group (Active Comparator): Patients in the IVC group will receive FOLFOX-based IVC combined with either cetuximab or bevacizumab every two weeks for a total of 8 weeks. The FOLFOX regimen consists of oxaliplatin (85 mg/m²) administered as a 2 hours intravenous infusion, leucovorin (400 mg/m²) administered as a 2 hours intravenous infusion, and fluorouracil (2400 mg/m²) administered as a 44 hours intravenous infusion, followed by intravenous administration of bevacizumab (5 mg/kg) or cetuximab (500 mg/m²).
  Cetuximab is used for the treatment of RAS/BRAF wild-type left-sided CRC, while bevacizumab is used for the treatment of RAS/BRAF wild-type right-sided CRC and RAS/BRAF mutant CRC regardless of tumor location.
  Interventions: Procedure: Intravenous Chemotherapy（IVC）

INTERVENTIONS:
Procedure: Transarterial infusion chemotherapy (TAIC) — TAIC can increase the local intra-tumoral concentrations of chemotherapeutic agents by intensifying drug delivery into the tumor via super-selective catheterization of the tumor-feeding artery, and meanwhile reduce systematic toxicity.
  Arms: TAIC Group
Procedure: Intravenous Chemotherapy（IVC） — Intravenous administration of chemotherapeutic agents is the mainstay of chemotherapy.
  Arms: IVC group

SUMMARY:
This is a prospective, multicenter, randomized, and open-label clinical trial. It is initiated to determine the efficacy of FOLFOX-based, transarterial infusion chemotherapy (TAIC) combined with either cetuximab or bevacizumab for patients with unresectable colorectal cancer (CRC).

DETAILED DESCRIPTION:
Current CRC treatment options include surgical resection, intravenous chemotherapy (IVC), radiation therapy, immunotherapy, and targeted therapy, or a combination of these options. IVC is an important therapy for CRC. Unfortunately, IVC results in broad drug distribution, while achieving with relatively low drug accumulation within the tumor. Compared with IVC, TAIC can increase the local intra-tumoral concentrations of chemotherapeutic agents by intensifying drug delivery into the tumor via super-selective catheterization of the tumor-feeding artery, and meanwhile reduce systematic toxicity. Hepatic artery infusion chemotherapy (HAIC) has been shown to yield significantly better outcomes than conventional transarterial chemoembolization (TACE) or IVC, and is now widely used for primary liver cancer and secondary liver malignancies. Based on these experiences, the investigators hypothesize that TAIC is clinically more effective at the same dose than IVC in the treatment of unresectable CRC. However, there is currently no high-quality evidence from clinical trials to support this hypothesis. To address this gap, the investigators will conduct a prospective study to verify this hypothesis. Eligible patients are those with unresectable CRC, those intolerant to surgical resection, and those with microsatellite instability or microsatellite instability low or proficient mismatch repair CRC. A total of 30 patients will be randomly assigned to the IVC group or TAIC group. Patients in the IVC group will receive the FOLFOX-based IVC with either cetuximab or bevacizumab every two weeks for a total of 8 weeks. Patients in the TAIC group will undergo FOLFOX-based TAIC combined with either cetuximab or bevacizumab on weeks 0 and 4 and will receive FOLFOX-based IVC with either cetuximab or bevacizumab on weeks 2 and 6. The primary endpoints are the objective response rate (ORR) and disease control rate (DCR).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Colorectal cancer confirmed by CT/MRI and colonoscopic biopsy；
3. Patients unfit for surgery due to poor general condition or tumor extent and location;
4. Patients who have not received prior chemotherapy or those who have undergone prior chemotherapy but remain chemosensitive.
5. Adequate haematological, heart, liver and renal functions are required, with the following specific criteria: white blood cell count≥4000/mL, neutrophils≥1500/mm³, platelets≥100×10⁹/L, haemoglobin≥10.0 g/L, total bilirubin 2.0 mg/dL, aspartate aminotransferase 100 IU/L, alanine aminotransferase 100 IU/L, serum creatinine 1.5 mg/dL or creatinine clearance rate≥60 mL/min/body, and urine protein/creatinine<1.
6. Patients have to have an expected life expectancy of ≥3months.
7. All the subjects in this study are required to sign an informed consent form.

Exclusion Criteria:

1. Patients with other primary malignant tumors;
2. Patients with gastrointestinal perforation;
3. Patients are allergic to the antitumor agents;
4. Women who are pregnant, breastfeeding, or planning to become pregnant;
5. Patients who receive other antitumor therapies concurrently, such as chemotherapy, targeted therapy, or radiotherapy;
6. Patients with MSI-H/dMMR CRC；
7. Patients for whom participation in the study is deemed to be inappropriate by the doctor in charge and/or the investigator for any other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 8 weeks
  ORR is defined as the percentage of complete response and partial response that is maintained for at least 4 weeks from the first radiological confirmation.
DCR | 8 weeks
  DCR is defined as the ORR plus the percentage of patients with stable disease.

SECONDARY OUTCOMES:
The change in level of carbohydrate antigen 199 | 8 weeks
The change in level of carcinoembryonic antigen | 8 weeks
The change in level of hemoglobin | 8 weeks
The change in level of nutritional status | 8 weeks
  Nutritional status is assessed based on the Inpatient Nutrition Risk Screening Scale 2002 (NRS2002). With a scoring range from 0 to 7 points, higher score indicates a more severe degree of malnutrition.
The change in level of frailty status | 8 weeks
  Frailty status is assessed based on the Clinical Frailty Scale (CFS). With a scoring range from 1 to 9 points, higher score indicates a more severe degree of frailty.
The change in level of performance status | 8 weeks
  Performance status is assessed based on the Eastern Cooperative Oncology Group (ECOG) score. With a scoring range from 0 to 5 points, a higher score indicates a poorer performance status.
Response rate of intestinal obstruction | 8 weeks
  Resolution of intestinal obstruction is defined as the subsidence of obstruction symptoms and signs, with the return of normal flatus and defecation.
The rate of conversion to resectable status | 8 weeks
  The assessment of surgical resectability by an experienced and dedicated multidisciplinary team is required at each tumor assessment.
R0 resection rate | 8 weeks
  The American Joint Committee on Cancer definition of R0 resection, any microscopically positive surgical margin on final pathologic review, is used.

OTHER OUTCOMES:
Adverse events | 8 weeks
  Adverse events are defined that newly appeared, increased in frequency, or worsened in severity following initiation of study drug. Adverse events were graded according to National Cancer Institute Common Terminology Criteria for Adverse Events, version 6.0.

CONTACTS AND LOCATIONS:
Overall Officials: Quanda Liu, MD, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Xicheng, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
At present, this study remains in the active implementation phase. Given that individual participant data (IPD) contains sensitive personal privacy information of research subjects, the investigators will not share the IPD with external researchers temporarily, in order to strictly comply with ethical requirements and fully protect the legitimate rights and interests of study participants.